CLINICAL TRIAL: NCT06684288
Title: Efficacy of Access Flap Surgery on Subgingival Periodontopathogen Levels in Periodontitis Patients: A Split-Mouth Randomized Clinical Trial
Brief Title: Efficacy of Access Flap Surgery on Subgingival Peridontopatgogens in Individuals With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ece AÇIKGÖZ ALPARSLAN, Assistant professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/80
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access flap surgery group (Experimental): Quadrants in participants requiring periodontal surgery were randomly assigned to access flap surgery sites. Following local anesthesia, a mucoperiosteal flap was elevated and handled with microsurgical instruments (blades, scalpel, needle holder, scissors, and tweezers; Carl Martin GmbH, Solingen, Germany) in accordance with the simplified papilla preservation flap (SPPF) technique.
  Interventions: Procedure: Access flap surgery
- Control group (No Intervention): untreated sites

INTERVENTIONS:
Procedure: Access flap surgery — Granulation tissue attached to the alveolar bone was excised to ensure complete access and optimal visibility of the root surfaces. In addition, instrumentation was performed using a combination of ultrasonic and hand instruments, and no alveolar bone modification was undertaken during the flap procedure. Subsequently, the mucoperiosteal flap was repositioned and primarily closed with proximal simple sutures employing monofilament suture material (5/0 Propilen, Dogsan, Türkiye). Patients were given post-operative recommendations; however, no medication was prescribed.
  Arms: Access flap surgery group

SUMMARY:
The participants in the present study were individuals diagnosed with stage III grade B periodontitis. Each patient underwent the first step of non-surgical periodontal treatment. In the first week following the initial session, the second step of the non-surgical periodontal treatment was performed on all four quadrants in a single appointment administered by the same blinded operator. Different sites of participating patients scheduled for periodontal surgery were assigned as either access flap surgery sites (test group) or untreated sites (control group) through a randomization procedure.

Each patient who met the study criteria underwent one of the following: one side of the mouth was treated with AFS, while the contralateral quadrants served as the control. All the access surgeries were conducted by the same blinded periodontist.

To evaluate the healing of periodontal tissues, detailed periodontal scores were recorded prior to and four weeks after access flap surgery.

The molecular genetic identification and quantification (qPCR) of subgingival periodontopathogens were performed by an operator who was blinded to group distribution. In the qPCR method, an increase in the number of cycles corresponds to a concomitant increase in the amount of DNA detected by the fluorescent dye. The Ct values obtained from the analysis results of subgingival plaque samples were integrated into the 2-ΔCt formula to calculate the difference in fold change occurring in the quantities of microorganisms.

Continuous variables were assessed for normality using the Shapiro-Wilk test. Subsequently, based on the normal distribution assumption, comparisons between independent groups were conducted using either the Student's t-test or the Mann-Whitney U test. For comparisons between dependent groups, the analyses employed either the Paired t-test or the Wilcoxon test.

DETAILED DESCRIPTION:
The participants in the present study were individuals diagnosed with stage III grade B periodontitis, as determined by the criteria established in the 2017 World Workshop for the Classification of Periodontal Diseases and Conditions.

Non-surgical periodontal treatment was administered to all quadrants in patients scheduled to participate in the study, using periodontal hand instruments (Gracey curettes, Hu-Friedy®; Chicago, IL) in conjunction with an ultrasonic device (Cavitron Plus, Dentsply®, Duisburg, Germany). Each patient underwent the first step of non-surgical periodontal treatment, which involved the mechanical removal of supragingival deposits, motivation, and personalized oral hygiene instructions, including interdental plaque control and toothbrushing using the modified Bass technique. In the first week following the initial session, the second step of the non-surgical periodontal treatment, which encompassed subgingival instrumentation (SI), was performed on all four quadrants in a single appointment administered by the same blinded operator. Patients did not receive any prescribed medication or mouthwash. At the one-month follow-up visit after SI (14 days pre-surgery), patients were clinically re-examined, and their compliance with the inclusion/exclusion criteria was reassessed. Patients requiring access flap surgery, indicated by the presence of deep residual pockets (PD ≥ 6 mm), were identified and underwent the randomization procedure. Different sites of participating patients scheduled for periodontal surgery were assigned as either access flap surgery sites (test group) or untreated sites (control group) through a randomization procedure. Other patients determined not to need access flap surgery were not included in the study and were instead enrolled in repeat subgingival instrumentation or a supportive periodontal care program.

Patients were assigned consecutive ascending numbers during the enrollment visit. Prior to the commencement of the study, the order of treatment quadrants was randomized by an investigator not directly involved in the examination or treatment process, using random sequences generated by a computer random-number generator. Allocation concealment was achieved using opaque sealed envelopes, sequentially numbered. Based on this process, the teeth on the right or left site were designated as the test group while those on the opposite site were assigned to the control group. The allocation remained concealed from the examiner throughout the periodontal examination and recordings, and the envelope was not opened by the operator until the first treatment visit.

Each patient who met the study criteria underwent one of the following: one side of the mouth was treated with AFS, while the contralateral quadrants served as the control. All the access surgeries were conducted by the same blinded periodontist Following local anesthesia, mucoperiosteal flap was elevated and handled with microsurgical instruments (Blades, scalpel, needle holder, scissor, and tweezer, Carl Martin GmbH, Solingen, Germany) in accordance with the simplified papilla preservation flap (SPFF) technique. Granulation tissue attached to the alveolar bone was excised to ensure complete access and optimal visibility of the root surfaces. In addition, instrumentation was performed using a combination of ultrasonic and hand instruments, and no alveolar bone modification was undertaken during the flap procedure. Subsequently, the mucoperiosteal flap was repositioned and primarily closed with proximal simple sutures employing monofilament suture material (5/0 Propilen, Dogsan, Türkiye). Patients were given post-operative recommendations; however, no medication was prescribed.

Periodontal measurements including probing depth (PD) (mm), clinical attachment level (CAL) (mm), bleeding on probing (BOP) (±), gingival index (GI), and plaque index (PI)were assessed at two distinct time intervals by a calibrated periodontist who was blinded to the experimental sites.20 These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed. To evaluate the healing of periodontal tissues, detailed periodontal scores were recorded prior to and four weeks after access flap surgery.

Among the periodontal scores recorded for each patient, four teeth (two for the treatment group and two for the control group) demonstrating the highest scores (PD ≥6 mm, CAL ≥5 mm) were designated as donor sites for subgingival plaque sampling. Sample collection was conducted before and one month after surgery by the investigator responsible for performing clinical measurements. Sampling sites were isolated using sterile cotton rolls, followed by the supragingival plaque removal from the tooth surface. Subsequently, sterilized paper points (Paperpoint #50, EndoPoint®, Paraiba do Sul, RJ, Brazil) were delicately inserted into the designated periodontal pockets, exerting gentle pressure until encountering mild resistance. The paper points were retained within the periodontal pocket for 20 seconds before being carefully transferred to sterile microcentrifuge tubes, securely capped for storage. The samples were stored in a -80°C freezer at Trakya University Technology Research and Development Application Center.

The molecular genetic identification and quantification of subgingival periodontopathogens were performed by an operator who was blinded to group distribution. The PureLink® Genomic DNA Mini Kit (INVITROGEN, Massachusetts, USA) was employed for DNA isolation. Samples within 1.5 ml centrifuge tubes were thawed at room temperature for dissolution after being retrieved from the -80°C freezer. DNA isolation proceeded according to the manufacturer's instructions, involving sequential steps of cell lysis, DNA binding to filter membranes, washing, and elution. Subsequently, the tubes containing the samples underwent centrifugation at 21,300 x g for 1 minute to procure pure genomic DNA of microorganisms. These isolated DNA samples were preserved at -20˚C until the PCR stage.

Within the Real-time quantitative PCR methodology, TaqMan® Probes (Applied Biosystems™, CA, USA) labeled with fluorochromes (fluorescent substances) at the 5' and 3' termini were utilized. The TaqMan Multiplex Master kit is a convenient pre-mixture of all components necessary, aside from primers and probes, to perform qPCR. It contains DNA polymerase, dNTPs (adenosine triphosphate, guanosine triphosphate, thymidine triphosphate, cytidine triphosphate), KCL or MgCL2, and polymerase buffer. The purpose of this technology is to detect known genomic, plasmid or complementary DNA (cDNA) sequences both qualitatively and quantitatively.

For PCR analyses, 20 μl of master mix (Applied Biosystems™, CA, USA) was placed in 96-well microplates. Then, 5 μl of the DNA sample taken from each case was added to some of these wells to serve as a test, while 5 μl of the sample taken from 3 healthy patients, which were not included in the study, was added to the remaining wells to serve as an internal control. These mixtures, each with a total volume of 25 μL, were run on the PCR machine (ABI 7500 Fast Real-Time PCR System, Applied Biosystems™, CA, USA) The qPCR study protocol included the following steps: a polymerase activation step (1 cycle at 95 °C for 3 min), a denaturation step (40 cycles at 95 °C for 15 s), and an annealing/extension step (40 cycles at 5 °C for 30 s).

In the context of the qPCR method, an increase in the number of cycles corresponds to a concomitant increase in the amount of DNA detected by the fluorescent dye. The threshold cycle value (Ct) refers to the cycle number at which the fluorescence radiation surpasses a predetermined threshold during amplification. In the present study, the Ct values obtained from the analysis results of subgingival plaque samples were integrated into the 2-ΔCt formula to calculate the difference in fold change occurring in the quantities of microorganisms.The disparity between the target bacteria detected at baseline and on the 1st month was computed utilizing the following formula:

ΔCt: [Ct_target bacteria in 1st month] - [Ct_target bacteria in baseline] The fold change in quantities of the target bacteria on 1st month compared to baseline: 2-Δ∆Ct All analyses were conducted using the SPSS version 23 software package (IBM Corp, Armonk, NY). Two groups, test and control, were defined with a substantial effect size (0.4) difference in microbial quantities and a significance level of 0.05. To assess correlations in repeated measurements with a correlation coefficient of 0.5, a sample size of 40 cases (20 test - 20 control) was determined using G*Power 3.1.9.2 software. The significance level was set at p < 0.05.

Continuous variables were assessed for normality using the Shapiro-Wilk test. Subsequently, based on the normal distribution assumption, comparisons between independent groups were conducted using either the Student's t-test or the Mann-Whitney U test. For comparisons between dependent groups, the analyses employed either the Paired t-test or the Wilcoxon test.

The correlation between continuous variables was investigated through Spearman correlation analysis. Continuous variables were described in terms of mean ± standard deviation (SD), median (interquartile range (IQR)), and range (minimum-maximum), while categorical variables were represented by frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Having 20 or more permanent teeth, excluding third molars and teeth with endodontic lesions;
* Exhibiting periodontitis with more than 30% loss of periodontal support tissue; - Having at least two non-adjacent teeth with a probing depth (PD) ≥6 mm, clinical attachment level (CAL) ≥5 mm, and radiographic bone loss extending to at least the middle of the root16;
* Presenting with bleeding on probing (BOP) in at least 40% of all periodontal sites17;
* Having at least one tooth per quadrant meeting the aforementioned PD and CAL criteria.

Exclusion Criteria:

* Pregnancy or lactation;
* Systemic diseases potentially affecting immune response (e.g., diabetes mellitus, bone metabolic diseases, HIV, immunosuppressive therapy, radiation);
* Presence of caries, restoration, or prosthesis adjacent to the sampling site;
* Use of anti-inflammatory drugs or antibiotics within the previous 3 months.

Ages: 36 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
The mean fold change in the quantities of P. gingivalis | Before and four weeks after surgery
  RT- qPCR was carried out to detect the 16S rRNA gene of subgingival red complex species. The mean fold change in P. gingivalis counts was analyzed.
The mean fold change in the quantities of T.denticola | Before and four weeks after surgery
  RT- qPCR was carried out to detect the 16S rRNA gene of subgingival red complex species. The mean fold change in T.denticola counts was analyzed.
The mean fold change in the quantities of T.forsythia | Before and four weeks after surgery
  RT- qPCR was carried out to detect the 16S rRNA gene of subgingival red complex species. The mean fold change in T.forsythia counts was analyzed.

SECONDARY OUTCOMES:
percentage of sites with BOP positive of each patient | Before and four weeks after surgery
  These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed
changes in the sum of the PI values of each patient | Before and four weeks after surgery
  These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed
changes in the sum of the GI values of each patient | Before and four weeks after surgery
  These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed
changes in mean PD values | Before and four weeks after surgery
  These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed
changes in mean CAL values | Before and four weeks after surgery
  These measurements were conducted on six different aspects of each tooth (disto-buccal/labial, mid-buccal/labial, mesio-buccal/labial, disto-lingual/palatinal, mid-lingual/palatinal, and mesio-lingual/palatinal) using a manual periodontal probe (Williams probe, Hu-Friedy®; Chicago, IL), and the average value was computed

CONTACTS AND LOCATIONS:
Overall Officials: Ece Açıkgöz Alparslan, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once the study results are converted into an article and published in a scientific journal, the study protocol may be shared. The authors will decide on this after the publication phase

REFERENCES:
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Coffey J, Choudhry M, Shlossman M, Makin IRS, Singh VK. Multiplex real-time PCR detection and relative quantification of periodontal pathogens. Clin Exp Dent Res. 2016 Aug 11;2(3):185-192. doi: 10.1002/cre2.37. eCollection 2016 Dec. PMID 29744166
- [Background] Kyriazis T, Gkrizioti S, Tsalikis L, Sakellari D, Deligianidis A, Konstantinidis A. Immunological and microbiological findings after the application of two periodontal surgical techniques: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Nov;40(11):1036-42. doi: 10.1111/jcpe.12149. Epub 2013 Aug 22. PMID 24033812
- [Background] Levy RM, Giannobile WV, Feres M, Haffajee AD, Smith C, Socransky SS. The effect of apically repositioned flap surgery on clinical parameters and the composition of the subgingival microbiota: 12-month data. Int J Periodontics Restorative Dent. 2002 Jun;22(3):209-19. PMID 12186343
- [Derived] Bayram C, Acikgoz-Alparslan E. Efficacy of Periodontal Surgery on Subgingival Periodontopathogen Levels in Periodontitis Patients: A Randomized Clinical Trial. Int J Dent. 2025 Dec 26;2025:4419048. doi: 10.1155/ijod/4419048. eCollection 2025. PMID 41476849